CLINICAL TRIAL: NCT04611776
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Adjuvant Platinum-Doublet Chemotherapy, With or Without Atezolizumab, in Patients Who Are ctDNA Positive After Complete Surgical Resection of Stage IB to Select IIIB Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Adjuvant Platinum-Doublet Chemotherapy, With or Without Atezolizumab, in Patients Who Are ctDNA Positive After Complete Surgical Resection of Stage IB to Select IIIB Non-Small Cell Lung Cancer
Acronym: CATHAYA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The positive results from IMpower010 demonstrated benefit by adding atezolizumab as adjuvant therapy in early stage NSCLC. These results raised ethical concerns of enrolling pts to best supportive care over checkpoint inhibition in this setting.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO41867
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Carboplatin; Cisplatin; Pemetrexed; Gemcitabine; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Atezolizumab + platinum-doublet followed by atezolizumab maintenance (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Paclitaxel
- Arm B: Placebo + platinum-doublet followed by placebo maintenance (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered intravenously during the induction phase and the maintenance phase.
  Other Names: Tecentriq
  Arms: Arm A: Atezolizumab + platinum-doublet followed by atezolizumab maintenance
Drug: Placebo — Placebo will be administered intravenously during the induction phase and the maintenance phase.
  Arms: Arm B: Placebo + platinum-doublet followed by placebo maintenance
Drug: Carboplatin — Carboplatin will be administered intravenously during the induction phase.
Drug: Cisplatin — Cisplatin will be administered intravenously during the induction phase.
Drug: Pemetrexed — Pemetrexed will be administered intravenously during the induction phase.
Drug: Gemcitabine — Gemcitabine will be administered intravenously during the induction phase.
Drug: Paclitaxel — Paclitaxel will be administered intravenously during the induction phase.

SUMMARY:
This is a Phase II, multicenter, double-blind, randomized study designed to evaluate the efficacy and safety of adjuvant treatment with atezolizumab in combination with platinum-doublet chemotherapy followed by atezolizumab compared with adjuvant placebo in combination with platinum-doublet chemotherapy followed by placebo in patients with Stage IB to IIIB (T3N2) NSCLC following surgical resection who are positive for ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Complete resection (R0) and pathologically confirmed Stage IB to select IIIB NSCLC (8th edition)
* Submission of pre-surgery blood sample and surgically resected tumor tissue slides or block
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Normal life expectancy excluding lung cancer mortality risk
* Positive ctDNA status in plasma confirmed by central laboratory testing after surgical resection and prior to start of adjuvant therapy.

Exclusion Criteria:

* Resected NSCLC with positive margins (R1 or R2)
* NSCLC with histology of large cell neuroendocrine carcinoma or sarcomatoid carcinoma
* Mixed NSCLC and SCLC histology
* Any prior therapy for lung cancer, including neoadjuvant therapy, or radiotherapy
* NSCLC with an activating EGFR mutation or ALK fusion oncogene
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2025-03-06 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
ctDNA Clearance Rate at 6 Months | Randomization up to 6 months
  ctDNA clearance rate at 6 months after randomization, defined as the proportion of participants with undetectable ctDNA at 6 months in the post-operative ctDNA+ participants.
Disease-Free Survival (DFS) | Randomization up to approximatly 159 months
  Disease-free survival (DFS), as assessed by the investigator, and defined as the time from randomization to the date of occurrence of any of the following, whichever occurs first: First documented local or distant recurrence of non-small cell lung cancer (NSCLC) after an integrated assessment of radiographic data, biopsy sample results (if available), and clinical status; Occurrence of new primary NSCLC (non-small cell lung cancer); Death from any cause in the post-operative ctDNA+ participants

SECONDARY OUTCOMES:
ctDNA Clearance Rate at 12 Months | Randomization up to 12 months
  ctDNA clearance rate in post-operative ctDNA+ participants.
Overall ctDNA Clearance Rate | Randomization up to approximately 159 months
  Overall ctDNA clearance rate in post-operative ctDNA+ participants.
Duration of ctDNA Clearance | Up to approximatly 159 months
  Duration of ctDNA clearance, defined as the time from the first documented ctDNA clearance to ctDNA detection, investigator-assessed radiographic or biopsy confirmed disease recurrence, or death from any cause, whichever occurs first in post-operative ctDNA+ participants.
Overall survival (OS) | Randomization to death from any cause (up to approximately 159 months)
  Overall survival (OS) after randomization, defined as the time from randomization to death from any cause in the post-operative ctDNA+ participants.
DFS Rate | Randomization to 2 years and 3 years
  DFS rate at 2 years and 3 years, defined as the probability that a participant has not experienced disease recurrence, a new primary NSCLC, or death from any cause, as determined by the investigator at 2 years and 3 years, respectively in the post-operative ctDNA+ participants.
Overall ctDNA Clearance Rate in the PD-L1 TC>=1% Population | Randomization up to approximately 159 months
  Overall ctDNA clearance rate in the PD-L1 TC>=1% (Ventana SP263) population in the post-operative ctDNA+ participants.
OS Rate | Randomization to 2 years and 3 years
  OS rate at 2 years and 3 years, defined as the probability that a patient has not experienced death from any cause at 2 years and 3 years, respectively in the post-operative ctDNA+ participants.
Time to Confirmed Deterioration (TTCD) in Patient-Reported Functioning and Global Health (GHS)/Quality of Life (QoL) | Up to approximately 159 months
  Time to confirmed deterioration (TTCD) in patient-reported functioning and global health (GHS)/quality of life (QoL), as measured by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30), and in patient-reported lung cancer symptoms for cough, dyspnea (a multi-item subscale), and chest pain, as measured through the use of the EORTC Quality-of-Life Questionnaire Lung Cancer Module (QLQ-LC13) in the post-operative ctDNA+ participants.
Percentage of Pariticipants with Adverse Events | Randomization up to approximatly 159 months
  Percentage of participants with adverse events in the post-operative ctDNA+ participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).